CLINICAL TRIAL: NCT03616080
Title: Effect of Soccer Play in Children With Cerebral Palsy
Brief Title: Soccer Play in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Bo Young Hong, Associate professor, The Catholic University of Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VC17ONSI0205
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: all were ambulatory children with CP age 5-12 years old.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): children who participated in soccer play program usual activity and therapy + soccer play program (once a week for eight weeks)
  Interventions: Behavioral: soccer play program
- control (No Intervention): children without soccer paly program usual activity and therapy

INTERVENTIONS:
Behavioral: soccer play program — once a week for an hour of a soccer program for 8 weeks
  Arms: experimental

SUMMARY:
1. To figure out the effect of soccer play (once a week for 8 weeks) on pulmonary function in children with cerebral palsy
2. To find out if the leisure activity (soccer) increase the quality of life, motor function, gait function etc..
3. Safety of soccer play in children with cerebral palsy

DETAILED DESCRIPTION:
1. 1 hr of play once a week for 8 weeks of soccer program was done in the experimental group.
2. Both the experimental and control group were children with ambulatory cerebral palsy aged 5 to 12 years.
3. Several outcomes were measured before and after the program

   * pulmonary function test including FVC, FEV1
   * GMFM-88, PBS, walking test, muscle power sprint test, timed up and go, gait parameters
   * Child Health Questionnaire Parent Form 50 (CHQ-PF50)
   * KIDSCREEN
4. An accelerometer was worn before the program and during the program for a week (experimental group only)

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy
* GMFCS level I-II
* 5-12 years old

Exclusion Criteria:

* acute disease, less than 6 months from the surgery
* the behavioral or psychiatric problem that hinders group activity
* intellectual disability to do the questionnaire
* who do not participate in the class well (absent more than 3 times)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change of FVC after soccer program | before and after the program, up to 10 weeks interval
  FVC, forced vital capacity (L)

SECONDARY OUTCOMES:
Change of gross motor function after soccer program | before and after the program, up to 10 weeks interval
  GMFM-88 (Gross motor function measure-88)
Change of balance after soccer program1 | before and after the program, up to 10 weeks interval
  Pediatric balance scale (PBS)
Change of balance after soccer program2 | before and after the program, up to 10 weeks interval
  timed up and go test (second)
Change of anaerobic test after soccer program | before and after the program, up to 10 weeks interval
  Muscle Power Sprint Test (MPST), Power (watt)
Change of physical activity with soccer program | before and during the program (about 3-4 weeks interval)
  wear an accelerometer for a week
Change of QOL (parents) | before and after the program, up to 10 weeks interval
  CHQ-PF50 (CHILD HEALTH QUESTIONNAIRE- PARENT FORM)
Change of QOL (children) | before and after the program, up to 10 weeks interval
  KIDSCREEN 27
Change of FEV1 after soccer program | before and after the program, up to 10 weeks interval
  FEV1, forced expiratory volume in 1 second (L)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Hong, Principal Investigator — St. Vincent's hospital, The Catholic University of Korea
Locations (1):
- St. Vincent's hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No